CLINICAL TRIAL: NCT00088712
Title: Event Related Potentials From Infancy to Adulthood
Brief Title: Event Related Potentials in Infants and Adults
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040250; 04-CH-0250
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-08-26

CONDITIONS: Healthy; Child Development
Keywords: Behavior and Neurocognition; Functional Brian Activity; Visual Perception; Selective Attention; Information Processing; Age Differences; Childhood Growth and Development; Cognitive Development; Brain Connectivity; Healthy Volunteer; HV
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

SUMMARY:
This study will explore the development of visual perception and the brain activity that underlies it. It will examine electrical activity in the brain while people are processing characteristics of the visual environment, and how that processing might change with development.

Infants who are within 2 weeks on either side of their 4-month birthday may be eligible for this study. A parent of the child also participates.

Parents who join the study are asked basic questions about their family, such as its size and ethnic make-up, their infant's birth date, complications of pregnancy or delivery, and any health problems of the infant, such as congenital developmental disorders or visual abnormalities.

Each family is seen at the clinic one time for a 45-minute visit. The infant is outfitted with an elastic net containing many small sensors that make contact with the scalp. He or she is then shown pictures on a computer screen. The sensors in the head net are connected to a computer that records the infant's brain activity while the infant watches the pictures on the screen. The head net is moistened with warm water before being applied, and is not uncomfortable to wear. Towels are available throughout the session to dry any excess moisture from the net.

DETAILED DESCRIPTION:
The major objective of this research is to better understand the response of the brain to significant stimulation in early and later development. The proposed work is designed to examine infants', children's, and adults' (especially mothers') responses to salient features of the external environment. To do so, the present research studies the biological bases and behavioral significance of natural preferences and information processing. The primary research strategy to be used consists of analyzing behavioral and brain responses to visual patterns. In a laboratory procedure, subjects will explore patterns and their brain electrical activity will be measured simultaneously with an electronic analysis system. In specific, five experiments of visual attention in human infants, and 1 experiment in adults are proposed. In the first experiment with infants, babies are hypothesized to look longer at more saturated colors; in a second experiment, babies are hypothesized to look longer at gratings aligned along the vertical and horizontal orthogonals than along the obliques. Because saturated colors and orthogonal stimulation elicit greater activity in visual system neurons and greater amplitude evoked potentials than desaturated colors or oblique stimulation, respectively, these two experiments explore the hypothesis that the simple visual stimuli to which infants preferably attend are those that are particularly appropriate in stimulating the geniculostriate or primary visual system. In the third experiment, we plan to trace the ontogeny of the mature brain response to whole patterns as opposed to parts of patterns. In a fourth experiment, we intend to compare region-specific activity when the surface features of a familiarized visual target change to that when its location changes. In the fifth experiment, we examine individual differences in the power metrics associated with attention to visual stimuli in relation to individual differences in their corresponding behavior coded by observers. In an experiment with children and adults we will explore brain responses and their localization in to pictures of familiar and unfamiliar faces.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be selected for inclusion in this study and each to follow on the basis of age, gestational status (i.e., full-term vs. pre-term birth), visual normality, and general health status. Once the recruitment letters have been mailed, a brief screening interview will be conducted with all parents who call to express an interest in participating. These parents will be asked about their infants birth date, expected due date, and any diagnoses of severe perinatal complications, visual abnormalities, and congenital developmental disorders. Infants with a gestational age of less than 36 weeks, and/or those with histories of severe perinatal complications, visual abnormalities, or a family history of color-vision deficiency will not be recruited for participation. Equal numbers of males and females will be recruited to participate.

Ages: 3 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 440 (Actual)
Dates: Start 2004-07-28; Study Completion 2019-08-26

PRIMARY OUTCOMES:
EEG response | Once following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Clay W. Mash, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] BERLYNE DE. The influence of the albedo and complexity of stimuli on visual fixation in the human infant. Br J Psychol. 1958 Nov;49(4):315-8. doi: 10.1111/j.2044-8295.1958.tb00669.x. No abstract available. PMID 13596573
- [Background] Bornstein MH, Arterberry ME, Mash C. Differentiated brain activity in response to faces of "own" versus "unfamiliar" babies in primipara mothers: an electrophysiological study. Dev Neuropsychol. 2013;38(6):365-85. doi: 10.1080/87565641.2013.804923. PMID 23971490
- [Background] Mash C, Bornstein MH, Arterberry ME. Brain dynamics in young infants' recognition of faces: EEG oscillatory activity in response to mother and stranger. Neuroreport. 2013 May 8;24(7):359-63. doi: 10.1097/WNR.0b013e32835f6828. PMID 23470433